CLINICAL TRIAL: NCT00004225
Title: Phase I Pilot Trial of Adenovirus p53 and Radiotherapy on Nonsmall Cell Lung Cancer
Brief Title: Gene Therapy Plus Radiation Therapy in Treating Patients With Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000067466; ECOG-8597
Record Dates: First submitted 2000-01-28; First posted 2003-01-27 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2004-04

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — advexin; Radiotherapy

INTERVENTIONS:
Biological: Ad5CMV-p53 gene
Radiation: radiation therapy

SUMMARY:
RATIONALE: Inserting the gene for p53 into a person's cancer cells may improve the body's ability to fight cancer. Radiation therapy uses high-energy x-rays to damage tumor cells.

PURPOSE: Phase I trial to study the effectiveness of gene therapy plus radiation therapy in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the feasibility and tolerability of adenovirus p53 gene therapy and radiotherapy in patients with non-small cell lung cancer with or without prior radiotherapy to the indicator lesion(s).
* Determine p53 and p21 expression and induction of apoptosis and necrosis in patients treated with this regimen.
* Assess any vector incorporation, antitumor response, local control, viral dissemination, and development of adenovirus antibodies in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients are stratified by prior radiotherapy to the indicator lesion(s) (yes vs no).

Adenovirus p53 is injected directly into an endobronchial lesion via bronchoscopy or into locoregional tumors via multiple percutaneous punctures under fluoroscopic, ultrasonic, or CT scan guidance on days 1, 3, and 8. Patients undergo radiotherapy beginning on day 2 and continuing for a total of 10 days.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven non-small cell lung cancer with at least 1 lesion accessible for endobronchial or percutaneous injection
* Measurable or evaluable disease
* Must have a requirement for palliative radiotherapy to the thorax
* Clinically stable enough to undergo 3 adenovirus injections

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0 or 1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Platelet count greater than 100,000/mm^3

Hepatic:

* PT and PTT normal

Renal:

* Not specified

Cardiovascular:

* No New York Heart Association class III or IV heart disease

Other:

* No active systemic viral, bacterial, or fungal infection requiring treatment
* No concurrent illness requiring hospitalization or IV medications or psychologic, familial, sociologic, geographic, or other concurrent condition that would preclude adequate follow up and compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior adenoviral gene therapy
* Any number of any type of other prior biologic therapy allowed

Chemotherapy:

* Any number of any type of prior chemotherapy allowed
* At least 2 weeks since prior systemic cancer therapy and no worse than grade 2 toxicity in any organ

Endocrine therapy:

* Any number of any type of prior endocrine therapy allowed

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy greater than 50 Gy if prior and concurrent radiation fields include the spinal cord
* No prior radiotherapy in fraction sizes greater than 2 Gy with the spinal cord in the concurrent radiation field

Surgery:

* At least 4 weeks since surgical resection of lung tissue
* At least 2 weeks since any other prior surgery requiring general anesthesia and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-01

CONTACTS AND LOCATIONS:
Overall Officials: Joan H. Schiller, MD, Study Chair — University of Wisconsin, Madison
Locations (1):
- Vanderbilt-Ingram Cancer Center at Vanderbilt Medical Center, Nashville, Tennessee, United States